CLINICAL TRIAL: NCT04493918
Title: Effectivity of Local Implantation of the Mesenchymal Stem Cell on Vertebral Bone Defect Due to Mycobaterium Tuberculosis Infection (Clinical Trial)
Brief Title: Effectivity of Mesenchymal Stem Cell on Vertebral Bone Defect Due to Mycobaterium Tuberculosis Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmad Jabir Rahyussalim (Other)
Responsible Party: Sponsor-Investigator, Ahmad Jabir Rahyussalim, Dr. dr. Rahyussalim SpOT(K), Indonesia University
Organization: Indonesia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-04-0389
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Spinal Tuberculosis; Mesenchymal Stem Cell
Keywords: Mycobacterium tuberculosis
MeSH Terms: conditions — Tuberculosis, Spinal | interventions — Sodium Chloride

STUDY DESIGN:
Masking Description: Participants do not know which treatment they receives. Outcome assessor is a radiologist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MSC Group (Experimental): Mesenchymal Stem Cell + NaCl 0,9% 2ml
  Interventions: Combination Product: Mesenchymal Stem cell + Nacl 0.9%; Combination Product: NaCl 0.9%

INTERVENTIONS:
Combination Product: Mesenchymal Stem cell + Nacl 0.9% — Patient who undergo surgery, debridement, decompression and posterior stabilization injection with Nacl 0.9% 2 ml + MSC 30 million unit
Combination Product: NaCl 0.9% — Patient who undergo surgery, debridement, decompression and posterior stabilization injection with Nacl 0.9% 2 ml

SUMMARY:
This study evaluates the effectiveness of locally implantation of mesenchymal stem cell on vertebral bone defects due to infection of mycobacterium tuberculosis. there are controlled participants who receives placebo and patients who receives implantation of MSc

DETAILED DESCRIPTION:
Mesenchymal Stem Cell are implanted in Spinal Tuberculosis patient. MSC has inflammatory effect and the ability to form into new bone.

In Spinal Tuberculosis, the spread of bacteria is commonly hematogenous, where the focus of infection is at the anterior part of the vertebrae near the subchondral bone. The infection process continues, where the necrotic casseous fragments formed into local abcess that may spread to the sorrounding area.

Patient with spinal tuberculosis who receives Anti TB Drug, is planned to undergo debridement, spinal stabilization. After thorough debridement, patient who fall into control group receives normal saline injection, patients who fall into treatment group will receive Mesenchymal Stem Cell.

ELIGIBILITY:
Inclusion Criteria:

* Clinicoradiologically diagnoses Spinal Tuberculosis
* receives Anti TB drugs
* minimun destruction 1/3 vertebral body

Exclusion Criteria:

* patient under 15 years old
* reject to be included in the study

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-21 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Vertebral bony fusion | 1 Year
  trabecular bone on xray and CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided